CLINICAL TRIAL: NCT00159900
Title: A Multicenter, Parallel Group Flexible Dose Study With A Double Blind, Randomized, Placebo Controlled Phase And An Open-Label Phase To Evaluate The Quality Of Erections In Men With Erectile Dysfunction Treated With Sildenafil Citrate
Brief Title: Quality of Erection Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481222
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate

SUMMARY:
The study objective is to evaluate the effect that sildenafil citrate has on the hardness of erections in males with erectile dysfunction, based on subject responses to question 5 on the Event Log (hardness of erection) as measured at the end of double blind treatment (week 6).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 18-55
* Documented clinical diagnosis of erectile dysfunction confirmed by an IIEF-EF Domain score of less than or equal to 25. (If the subject scores greater than 25 on the IIEF-EF Domain, screening procedures should be terminated.)

Exclusion Criteria:

* Subjects who have been treated with more than 6 doses of sildenafil citrate or any other phosphodiesterase type 5 (PDE-5) inhibitor such as vardenafil or tadalafil for erectile dysfunction [Note: subjects should not have taken any PDE-5 inhibitors within 4 weeks prior to the date of screening]

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 2005-05; Study Completion 2006-01

PRIMARY OUTCOMES:
Responses to Question 5 (erectile hardness) of the Event Log as measured from baseline to the end of double-blind treatment (week 6).

SECONDARY OUTCOMES:
Responses to the Quality of Erectile Questionnaire (QEQ) Responses to International Index of Erectile Function (IIEF) Domains (Erectile Function; Orgasmic Function; Sexual Desire; Intercourse Satisfaction; Overall Satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Brazil (4):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Rio Claro, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Germany (5):
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Rosenheim
  - Pfizer Investigational Site, Starnberg
- Italy (3):
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Roma
- Poland (4):
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Szczecin
  - Pfizer Investigational Site, Warsaw
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Bursa
  - Pfizer Investigational Site, Diyarbakır
  - Pfizer Investigational Site, Istanbul
  - Pfizer Investigational Site, Izmir

REFERENCES:
- [Derived] Kaminetsky JC, Stecher V, Tseng LJ. Quality of erections by age group in men with erectile dysfunction. Int J Clin Pract. 2017 Oct;71(10). doi: 10.1111/ijcp.12976. Epub 2017 Sep 11. PMID 28892218